CLINICAL TRIAL: NCT00295737
Title: 05/04 IMHOTEP-1 FHG: Ex Vivo Effect of an Immunotoxin on Activated Human Macrophages From Atopics After Segmental Instillation of Allergen and Endotoxin
Brief Title: Effect of an Immunotoxin on Activated Human Macrophages in Those With Allergic Rhinitis or Mild Intermittent Asthma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: proof of mechanism achieved with fewer subjects than anticipated
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 05/04 IMHOTEP-1 FHG
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Atopy; Rhinitis; Bronchial Asthma
Keywords: allergic rhinitis
MeSH Terms: conditions — Rhinitis; Asthma; Rhinitis, Allergic | interventions — Bronchoscopy; Allergens

INTERVENTIONS:
Procedure: bronchoscopy, allergen/endotoxin instillation

SUMMARY:
The primary objective of this study is to isolate macrophages by using bronchoalveolar lavage (BAL) for different in vitro experiments.

Therefore, following a baseline BAL, allergen, endotoxin, and saline will be instilled into three different lung segments during the first bronchoscopy. After 24 hours during a second bronchoscopy, BAL fluid will be collected in these challenged segments to harvest invaded cells for in vitro experimentation. In addition, segmental bronchial biopsies will be taken to assess the degree of local inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of atopy (allergic rhinitis or mild intermittent asthma)
* Age 18-55 years
* Nonsmoker (> 5 years)
* Forced expiratory volume in 1 second (FEV1) > 70% of the predicted value
* A positive skin prick test for grass mix or D. pteronyssinus at or within 12 months prior to the screening visit
* Informed consent
* Females with negative pregnancy test

Exclusion Criteria:

* Infections of the respiratory tract within the last month
* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
* Pathological findings in blood tests (differential blood count, blood clotting, electrolytes, liver enzymes, retention parameters)
* Subject is undergoing allergen desensitization therapy
* Permanent medication
* Systemic or inhaled corticosteroid use within the last month
* Anti-inflammatory medication within the last month
* Pregnancy
* Neurological or psychiatric disease or history of drug or alcohol abuse which would interfere with the subject's proper completion of the protocol assignment
* There is a risk of non-compliance with study procedures
* Participation in a clinical trial 30 days prior to enrolment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2006-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
number of macrophages in bronchoalveolar lavage | one day after challenge

SECONDARY OUTCOMES:
number of other BAL cells | one day after challenge

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hohlfeld, MD, Principal Investigator — Fraunhofer ITEM
Locations (1):
- Fraunhofer ITEM, Hanover, Germany